CLINICAL TRIAL: NCT06446635
Title: Semiflex Assisted Vacuum Therapy for Perianal Abscesses/Sinuses and Fistula: a Pilot Study
Acronym: Semiflex Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81105
Record Dates: First submitted 2024-05-06; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Perianal Fistula; Perianal Fistula Due to Crohn's Disease; Perianal Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a perianal abscess/sinus (Experimental)
  Interventions: Device: Semiflex Dome Catheter System
- Patients with perianal fistula (Experimental)
  Interventions: Device: Semiflex Dome Catheter System

INTERVENTIONS:
Device: Semiflex Dome Catheter System — Abces: In patients that present with a perianal abscess/sinus the semiflex dome catheter is inserted under general anesthesia. A small cut is made to drain and irrigate the septic sinus.
  Fistula: Under general anesthesia the seton is removed, the internal opening is excised and the internal opening is closed with a 2-0 Vicryl cross stitch.
  Both: Before surgery, the length of the tract is measured on MRI or CT. A Semiflex Catheter with the appropriate length and a diameter is selected. If during surgery appears that this is not the appropriate size, a different size catheter can be used. The catheter is fixed on a Renasys Adhesive gel patch (Smith and Nephew). The catheter is connected with a tubing system to a vacuum pomp with an average vacuum pressure of 80 cm H2O. The tube will be taped on the patient. After every 2-3 days the catheter will be exchanged by a 3-6 mm shorter catheter.

SUMMARY:
Rationale: Perianal fistulas are a common, invalidating problem for which a more effective and widely applicable treatment is necessary. Vacuum therapy has become one of the main pillars for management of a wide variety of (chronic) wound healing problems. A novel catheter set was developed for vacuum therapy of perianal abscesses/sinuses and fistulas: The Semiflex Dome System. This system will allow for a better and faster treatment and it will offer conformability with various fistula shapes and sizes.

Objective: With this pilot study, the investigators aim to test our novel catheter set for vacuum therapy of perianal abscesses/sinuses and fistulas for feasibility and efficacy.

Study design: The design of this prospective, multicentre study is a feasibility study.

Study population: Patients (≥ 18 years) with (Crohn's) perianal fistulas and patients with perianal abscesses/sinuses are eligible.

Intervention: A tailored (length and diameter) Semiflex dome catheter is inserted under general anaesthesia, after 6 weeks of seton drainage in patients with a perianal fistula and right away in patients with a perianal abscess/sinus. The catheter is fixed on a Renasys Adhesive gel patch (Smith and Nephew) and is connected with a tubing system to a vacuum pomp with an average vacuum pressure of 80 cm H2O. After two - three days the catheter will be exchanged by a shorter catheter in the outpatient setting. The therapy is continued for a maximum of four weeks in patients with a perianal abscess/sinus and two weeks in patients with perianal fistulas.

Main study parameters/endpoints: The primary objective of the study is the feasibility of the methodology with respect to smoothness of insertion and changing the semiflex catheters, capability of proper fixation of the catheter and maintaining vacuum for more than 48 hours, and compliance to the therapy in terms of pain and discomfort. Secondary objectives are efficacy of drainage of the perianal abscess/sinus, efficacy of curing the perianal abscess/sinus in terms of complete collapse of the sinus and disappearance of induration, efficacy of management of perianal fistula in terms of clinical and radiological healing, and safety in terms of complications.

Nature and extent of the burden and risks associated with participation: The Semiflex Dome Catheter System will be placed in patients with perianal fistulas and perianal abscess/sinus who would otherwise be treated using prior-art passive drainage catheters or repurposed vacuum-assisted closure therapy sponges. There are no known additional risks stemming from the proposed therapy. The Semiflex Dome Catheter System is made entirely of medical-grade silicone certified with ISO 10993- 05 and ISO 10993-10. The catheters will be connected with a tube configured to be connected to a CE certified vacuum generating system.

Sample size: Since this is a pilot study no sample size is required. The pilot study will consist of 2 parts. In the first part, 10 patients in each study group will be included and it will be assessed per study group if the catheter meets the proof of principle. After a positive result in one or both study groups, the second part of the study will start. 10 patients in each study group will be included. The proposed treatment protocol is considered feasible if at least 70% of the Semiflex dome catheter treatment per study group meets the four primary objectives.

ELIGIBILITY:
Inclusion criteria

* Perianal abscess/sinus or (Crohn's) perianal fistula
* ≥ 18 years and < 80 years
* Written informed consent

Exclusion criteria

* Patients with more than 2 external perianal openings
* Rectovaginal fistula
* Life expectancy < 2 years
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Smoothness of insertion and exchanging of the Semiflex catheter | 3 months
  The doctor will determine how easy the catheter is to insert on a scale of 0-10, with 0 being very difficult and 10 being very easy. A score <5 is considered as not smooth. This will be scored individually and if all primary outcome measures are met, the treatment is considered successful in this participant.
Proper fixation of the Semiflex catheter | 48 hours
  The system is properly fixed if it has been in place for >48 hours. If the system becomes loose before 48 hours, it is considered as not properly fixed. This will be scored individually and if all primary outcome measures are met, the treatment is considered successful in this participant.
Maintaining vacuum for more than 48 hours | 48 hours
  The system is properly vaccuum if it has been vacuum for >48 hours. If the system looses vaccuum before 48 hours, it is considered as not properly vaccuum. This will be scored individually and if all primary outcome measures are met, the treatment is considered successful in this participant.
Compliance to the therapy in terms of pain and discomfort | 3 months
  The patient gives a painscore after the Semiflex exchange on a scale of 0-10, with 0 being not painfull and 10 being very painfull. A score >5 is considered as too painfull. This will be scored individually and if all primary outcome measures are met, the treatment is considered successful in this participant.

SECONDARY OUTCOMES:
Efficacy of drainage of the perianal abscess/sinus | 3 months
  Is the Semiflex capable of draining the perianal abcess/sinus. 1 month after therapy a clinical evaluation will be done to see if the perianal abscess/ sinus is healed. Clinical closure is defined as closure of the external opening without discharge of pus on palpation. After three months a MRI is made to see if the perianal abscess/sinus is radiological healed. Radiological healing defined as complete fibrosis of the abscess/sinus on MRI.
Efficacy of management of perianal fistula in terms of clinical and radiological healing | 3 months
  Is the Semiflex capable of draining the perianal fistula. 1 month after therapy a clinical evaluation will be done to see if the perianal fistula is healed. Clinical closure is defined as closure of the external opening without discharge of pus or feaces on palpation. After three months a MRI is made to see if the perianal fistula is radiological healed. Radiological healing defined as complete fibrosis of the perianal fistual.
Safety in terms of complications | 3 months
  All complications related to the Semiflex treatment will be recorded during the follow-up of three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No